CLINICAL TRIAL: NCT01389466
Title: Randomized Phase I/II Study to Evaluate the Safety and Immunogenicity of 'MG1109(Egg-based, Pre-pandemic Influenza(H5N1) Vaccine)' Administered Intramuscularly in Healthy Adult Volunteers
Brief Title: Study to Evaluate the Safety and Immunogenicity of MG1109 in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Green Cross Corporation (Industry)
Collaborators: Korean Center for Disease Control and Prevention (Other Government)
Responsible Party: Sponsor
Organization: GC Biopharma Corp (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MG1109_P1/2
Record Dates: First submitted 2011-06-19; First posted 2011-07-08 (Estimated); Last update posted 2014-11-21 (Estimated); Status verified 2014-11

CONDITIONS: Influenza
Keywords: Avian influenza
MeSH Terms: conditions — Influenza, Human; Influenza in Birds | interventions — SE 1-step Futurabond M

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- MG1109 - Step 1 (Experimental)
  Interventions: Biological: Step 1
- Normal Saline - Step 1 (Placebo Comparator)
  Interventions: Biological: Step 1
- MG1109 - Step 2 (Experimental)
  Interventions: Biological: Step 2

INTERVENTIONS:
Biological: Step 1 — Investigational Product : MG1109 Dose : Cohort 1 : 0.125 mL Cohort 2 :0.25 mL Cohort 3 :0.5 mL Cohort 4 :1.0 mL intramuscularly injection, twice at an interval of 21 days
  Arms: MG1109 - Step 1; Normal Saline - Step 1
Biological: Step 2 — Investigational Product : MG1109 Dose : Cohort 1 :0.5 mL Cohort 2 :1.0 mL intramuscularly injection, twice at an interval of 21 days
  Arms: MG1109 - Step 2

SUMMARY:
This study was designed in two steps with Step 1, a single-center, double-blind, randomized clinical Pilot study and Step 2, a multi-center, single-blind, randomized clinical Pivotal study. The investigator evaluate the immunogenicity and safety of the investigational vaccine in the subjects during their participation in the study.

DETAILED DESCRIPTION:
MG1109 is purified, inactivated influenza viral antigen.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults who are available for follow-up during the study

Exclusion Criteria:

* Subjects with history of exposure to the H5N1 subtype or H5N1 subtype vaccine
* Subjects with immune system disorder including immune deficiency disease

Ages: 18 Years to 58 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 346 (Actual)
Dates: Start 2010-02; Primary Completion 2011-11 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects achieving post-vaccination Hemagglutination Inhibition(HI) antibody titer ≥ 1:40 in each dose group | 42 days after vaccination
Number of subjects with Solicited / Unsolicited adverse events | With in 24 weeks after vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Woo Joo Kim, MD, Ph.D, Principal Investigator — Korea University Guro Hospital
Locations (4):
- South Korea (4):
  - Korea University Ansan Hospital, Ansan
  - Inha University Hospital, Inchon
  - Korea University Guro Hospital, Seoul
  - Catholic University Of Korea ST. Vincent's Hospital, Suwon